CLINICAL TRIAL: NCT03331003
Title: "iRestore" Light Therapy Apparatus in the Treatment of Androgenetic Alopecia: A Randomized, Double-blind, Self-comparison, Sham Device-controlled, Multicenter Trial
Brief Title: "iRestore" Light Therapy Apparatus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201310067DSB
Record Dates: First submitted 2017-10-18; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2014-03

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low level light therapy (Experimental): 1 group uses the investigational device on the left side, and the subjects will have half part receiving low level light therapy (red light-emitting diode and laser irradiation)
  Interventions: Device: low level light therapy
- non-LLLT wavelength group group (Placebo Comparator): the control device on the right side, other half with non-low-level laser therapy wavelength (white light-emitting diode light bulb coating with red paint to make the irradiating light close to the red).
  Interventions: Device: non-LLLT wavelength group

INTERVENTIONS:
Device: low level light therapy — iRestore low-level light therapy on androgenetic alopecia
  Arms: low level light therapy
Device: non-LLLT wavelength group — A LED light device is non-curative for the patients.
  Arms: non-LLLT wavelength group group

SUMMARY:
Current effective therapies of pattern hiar loss are topical minoxidil and oral finasteride. Finasteride is an inhibitor of type 2 5α-reductase and will cause hypospadias in male infant if taken or touched by pregnant woman. The effect of minoxidil is still known now but the dilation of scalp vessel might improve the progression of pattern hair oss. However, minoxidil is not effective for frontotemporal recession and sometimes cause scalp irritation.

Low-level laser therapy (LLLT) a new therapy to treat alopecia. In 2007, LLLT was approved by the FDA as a treatment for hair loss. In some small studies, patients had a decrease in the number of vellus hairs, an increase in the number of terminal hairs, and an increase in shaft diameter. Up to now, however, no longer, placebo-controlled studies have proved its efficacy in this application.

According to the mechanism of paradoxical hair growth (PHG), sublethal injury to the hair follicle could stimulate the hair follicle to enter anagen via the release of factors that alter angiogenesis, leading to increased blood flow to the dermal papilla. Furthermore, load inflammation in the papilla nad heat shok response, possibly mediated by HSP27, may play a role in activation of follicular stem cell.

This study is a randomized, blinded, self-comparison and superior clinical trial design. In this clinical trial, the investigators try to evaluate the efficacy of low-level laser therapy in treating pattern hair loss. Pattern hair loss is characterized by increased vellus hairs and decreased shaft diameter, and these features are improved by LLLT in previous.

DETAILED DESCRIPTION:
This study is A randomized, double-blind, self-comparison, sham device- controlled, multicenter Trial. Total subjects is 100 and the clinical trial was conducted in National Taiwan University Hospital and National Taiwan University Hospital-Hsinchu Branch. The study starts from December 2013 to June 2015 for within 18 months.

The potential subjects will be collected into the clinical study, and have 24 weeks of treatment. The forth, twelve and twenty-fourth weeks are took as evaluation point. Besides the photo shooting area, recording the density of hair growth, analyzing of hair growth number, and the width of hair will be quantified. At the same time, the subject will also have the safety evaluation to see if there are any reddish or skin disorder(erythema, edema, dried, skin keratinization) or other systematic symptom. After quantifying the data, the degree of covered area in target area is seen as primary end point.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects of either gender who are 25-60 years old.
2. The male-pattern alopecia in men belongs to Stages IIa-V of the Norwood-Hamilton Scale;
3. The male-pattern alopecia in women belongs to Stages I-4, II-1 and II-2 of the Ludwig (Savin) Scale.
4. The subjects shall agree to have temporary punctate tattoo at the observed part.
5. There was continuous hair loss during the past 12 months.
6. Women with fertility shall agree to adopt appropriate contraception measures, including the intrauterine device, condom, spermicide, abstinence, vasoligation of the sexual partner, etc.
7. The skin type ranges between Types I and IV of Fitzpatrick scale, as shown in Table 1.
8. The subjects agree to shave off the hair at the observed part.
9. The photographic release form shall be read carefully before the signature.
10. The informed consent form shall be read carefully to understand the detailed trial content and the signature shall be made without any disturbance.

    * Table 1. Fitzpatrick Skin Typing

      * Always burns, never tans
      * Usually burns, tans minimally
      * Frequently burns and tans (light brown)
      * Rarely burns, tans easily (brown)
      * Very rarely burns, tans very easily (brown)
      * Never burns (dark brown to black)

Exclusion Criteria:

1. Use or administration of the following drugs within 6 months before the recruitment:

   * Minoxidil, finasteride or other inhibitors of 5α-reductase;
   * The drugs that may inhibit androgen, such as cyproterone, spironolactone, ketoconazole, flutamide and bicalutamide.
   * The drugs that may cause hirsutism, such as ciclosporin, diazoxide, phenytoin, Propecia, Dutasteride and psoralens, or other drugs for treating prostatic hypertrophy.
   * Oral adrenal corticoid (except inhaler adrenal corticoid)
   * The drugs with possible phototoxicity, such as tetracyclins, thiazides and certain NSAIDS.
   * Lithium or antischizophrenic drugs (phenothiazines);
   * Any drugs that will influence the assessment results or subjects' safety according to the opinions of the principal investigator.
   * Anti-cancer drugs.
2. Pregnant or breastfeeding women or those plan to get pregnant during the trial. The women with fertility shall take the contraceptive drugs orally or have the implantation, injection or subcutaneous injection of contraceptive drugs.
3. Patients with Type 2 diabetes.
4. Patients with heart disease who take phototoxic drugs.
5. Those who don't agree to maintain the hairstyle and hair color during the trial.
6. Those who had hair transplantation, scalp reconstruction procedure, hair braiding or scalp tattoo, which will influence the assessment results of the test or the subjects' safety according to the opinions of the principal investigator.
7. Those who use or once used depilation agents, laser hair removal or beeswax on the scalp to remove the hair or perform any action which will influence the assessment results of the trial according to the opinions of the principal investigator.
8. There is psoriasis, dermatitis, eczema or severe acne on the scalp.
9. Those who suffer from the diseases which may influence the hair growth according to the opinions of the principal investigator, such as the immunodeficiency syndrome, connective tissue-related diseases or infectious baldness.
10. Those with insignificant contrast of scalp and hair color, such as light skin color or white hair.
11. Inability to cooperate with the trial: those subjects who can't use the device or pay a return visit periodically according to the instruction of the physician or hospital during the trial in the opinions of the principal investigator.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Hair coverage of the targeted area | In the 24th week
  The photomicrography is taken to record the hair growth in the target area. The Folliscope (IBS-01 Pro Beauty Scope, Kowa Optics Corp.) is used to record the hair coverage in the tattooed area and analyze the hair growth number. The photography of the global scalp is also taken to record the top scalp and hair line shapes of the subjects. Hair coverage equals to ∑_(i=1)^n*π R_i^2

SECONDARY OUTCOMES:
evaluate the hair coverage | in the 4th and 12th weeks
  The Paired-T or McNemar's test is adopted to evaluate the hair coverage in the 4th and 12th weeks.
evaluate the increased hair thickness of the targeted area | in the 4th, 12th and 24th weeks
  The Paired-T test is adopted to evaluate the increased hair thickness of the targeted area
number of the hair in the targeted area | in the 4th, 12th and 24th weeks
  The Paired-T test is adopted to evaluate the number of the hair in the targeted area.
global assessment of the hair growth condition | in the 4th, 12th and 24th weeks
  The principal investigator will carry out the global assessment of the hair growth condition. The Wilcoxon rank sum test is adopted for comparison and the line chart is used to demonstrate the trend of the treatment effect. The scores of global assessment of the hair growth condition is 1, and 1 refers to thin.
global assessment of the hair growth condition | in the 4th, 12th and 24th weeks
  The principal investigator will carry out the global assessment of the hair growth condition. The Wilcoxon rank sum test is adopted for comparison and the line chart is used to demonstrate the trend of the treatment effect. The scores of global assessment of the hair growth condition is 3, and three refers to dense.
global assessment of the hair growth condition | in the 4th, 12th and 24th weeks
  The principal investigator will carry out the global assessment of the hair growth condition. The Wilcoxon rank sum test is adopted for comparison and the line chart is used to demonstrate the trend of the treatment effect. The scores of global assessment of the hair growth condition is 2, and 2 refers to medium, and three refers to dense.
global assessment of the hair growth condition | in the 4th, 12th and 24th weeks
  The principal investigator will carry out the global assessment of the hair growth condition. The Wilcoxon rank sum test is adopted for comparison and the line chart is used to demonstrate the trend of the treatment effect. The scores of global assessment of the hair growth condition is 0, and 0 refers to no hair growth.
The subjects' overall satisfaction assessment | in the 4th, 12th and 24th weeks
  The subjects' overall satisfaction assessment shall be carried out. The Wilcoxon rank sum test is adopted for comparison and the line chart is used to demonstrate the trend of the treatment effect.
  The scores of subject's satisfaction is 0 refers to dissatisfy.
The subjects' overall satisfaction assessment | in the 4th, 12th and 24th weeks
  The subjects' overall satisfaction assessment shall be carried out. The Wilcoxon rank sum test is adopted for comparison and the line chart is used to demonstrate the trend of the treatment effect.
  The scores of subject's satisfaction is 1 that refers to slightly satisfy.
The subjects' overall satisfaction assessment | in the 4th, 12th and 24th weeks
  The subjects' overall satisfaction assessment shall be carried out. The Wilcoxon rank sum test is adopted for comparison and the line chart is used to demonstrate the trend of the treatment effect.
  The scores of subject's satisfaction is 2 that refers to moderately satisfy.
The subjects' overall satisfaction assessment | in the 4th, 12th and 24th weeks
  The subjects' overall satisfaction assessment shall be carried out. The Wilcoxon rank sum test is adopted for comparison and the line chart is used to demonstrate the trend of the treatment effect.
  The scores of subject's satisfaction is 3 that refers to satisfy.
The subjects' overall satisfaction assessment | in the 4th, 12th and 24th weeks
  The subjects' overall satisfaction assessment shall be carried out. The Wilcoxon rank sum test is adopted for comparison and the line chart is used to demonstrate the trend of the treatment effect.
  The scores of subject's satisfaction is 4 that refers to Highly satisfy.